CLINICAL TRIAL: NCT04780906
Title: Influence of Wrist Taping on Handgrip Strength in Crossfit Athletes - Crossover Randomized Controlled Trial
Brief Title: Influence of Wrist Taping on Handgrip Strength in Crossfit Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vita Care (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 103
Record Dates: First submitted 2021-02-23; First posted 2021-03-04 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Sport Injury; Hand Injury Wrist
Keywords: sports

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham first (group 1) (Sham Comparator): Performs the first round of test with the sham comparator than with the experimental wrist taping
  Interventions: Other: Wrist taping
- Wrist taping first (group 2) (Experimental): Performs the first round of test with the experimental wrist taping than with the sham comparator
  Interventions: Other: Wrist taping

INTERVENTIONS:
Other: Wrist taping — Wrist taping as used as standard in CrossFit practice

SUMMARY:
The idea that the use of a wristband can increase the grip strength is old, but without systematic scientific evidence. Most Crossfit practitioners wear wrist bands during training because it is believed that the wristband increases the grip strength of the hand. The aim of this study is to to analyze the influence of the use of the wristband on the maximum force value and on the dynamic resistance of hand hold. A simple blind randomized cross-over trial will be performed.

ELIGIBILITY:
Inclusion Criteria:

* be an amateur practitioner of the Crossfit modality with at least 6 months of regular sports practice (at least 4 times a week)
* between 18-40 years old
* agree to participate in the study and sign the informed consent form (ICF).

Exclusion Criteria:

* active wrist/ arm injury or pain on the day of the test (pain score greater than 3 in 10 for both shoulder, forearm, wrist and / or hand on the VAS pain scale)
* history of wrist injury (especially fracture or ligament injury)
* previous wrist surgery

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Grip | 0 minutes; 5 minutes
  Mean of the first 3 hand pressures (kg) measured by hand dynamometer

SECONDARY OUTCOMES:
Endurance | 0 minutes; 5 minutes
  Percentage (%) of strength measured in the last 3 movements in relation to the first 3 movements

CONTACTS AND LOCATIONS:
Overall Officials: Luis Marchi, PhD, Study Director — Instituto Vita
Locations (1):
- Instituto Vita, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No